CLINICAL TRIAL: NCT01368861
Title: Effective Analgesia Using the 5 S's During Routine Immunizations at 2 and 4 Months
Brief Title: Effective Analgesia During Routine Immunizations
Status: Completed | Type: Observational
Sponsor: Children's Hospital of The King's Daughters (Other)
Responsible Party: Principal Investigator, John Harrington, Associate Professor, Children's Hospital of The King's Daughters
Other Study IDs: EVMS
Record Dates: First submitted 2011-06-03; First posted 2011-06-08 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Pain
Keywords: infant; immunizations; pain; pain management; vaccines; analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- control: water and normal physical comfort provided by mom
- sucrose: sugar and normal physical comfort provided by mom
- physical intervention: physical intervention using the 5 S's and water
- physical intervention and sucrose: Physical intervention using the 5 S's and sugar water

SUMMARY:
The purpose of this study is to observe and measure the analgesic effectiveness of the 5 S's (swaddling, side/stomach position, shushing, swinging, and sucking) alone and combined with sucrose, during routine immunizations at 2 and 4 month well child visits.

DETAILED DESCRIPTION:
Study Procedure

Infants meeting inclusion criteria were identified daily by reviewing the list of patients scheduled for a 2 or 4 month well child visit at the outpatient site. The parent or legal guardian was approached prior to vaccination by the research assistant for participation in the study. If the parent/guardian accepted to participate in the vaccine study, the consenting process was performed and patients were brought to a designated examination room. Infants of parents or guardians who consented were randomly assigned to one of four study groups using pre-sealed cards. Ten cards were assigned to each group for a total of 40 cards, which were recycled with each group of 40 infants enrolled into the study. The four groups of the study included:

1. 2 ml of water 2 minutes prior to immunization and comfort by parent or guardian after Immunization (Control Group)
2. 2 ml of 24% oral sucrose 2 minutes prior to immunization and comfort by parent or guardian after immunization (Sucrose Group)
3. 2 ml of water 2 minutes prior to immunization and physical intervention using the 5 S's by researcher after immunization (Physical Group)
4. 2 ml of 24% oral sucrose 2 minutes prior to immunization and physical intervention using the 5 S's by researcher after immunization (Physical and Sucrose Group)

ELIGIBILITY:
Inclusion Criteria:

* infants with a gestational age between 32-42 weeks at delivery and post-natal age of less than 20 weeks old

Exclusion Criteria:

* acetaminophen or ibuprofen administration within 4 hours prior to immunization, current neurological disorder, known genetic anomaly, moderate to severe illness with or without fever at the time of vaccination, anaphylactic reaction to previous dose of vaccine, or if infant was previously enrolled in the study at 2 months.

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All patients were enrolled from the General Academic Pediatric outpatient practice located at The Children's Hospital of The King's Daughters in Norfolk, VA. This practice serves a predominantly urban, Medicaid enrolled, African-American population and has approximately 30,000 annual visits per year.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To measure analgesic effectiveness of the 5 S's (swaddling, side/stomach position, shushing, swinging, and sucking) alone and combined with sucrose, during routine immunizations at 2 and 4 month well child visits. | every 15 sec
  Does the 5 S's improve the percieved pain of infants receiving vaccinations. The Modified Riley Pain Scale which measure 3 aspects of pain was utilized. The scale is validated for the assessment of acute pain in preterm and term infants.

CONTACTS AND LOCATIONS:
Overall Officials: John W Harrington, MD, Principal Investigator — Children's Hospital of The King's Daughters
Locations (1):
- Children's Hospital of The King's Daughters, Norfolk, Virginia, United States

REFERENCES:
- [Background] Ornstein PA, Manning EL, Pelphrey KA. Children's memory for pain. J Dev Behav Pediatr. 1999 Aug;20(4):262-77. doi: 10.1097/00004703-199908000-00009. PMID 10475601
- [Background] Taddio A, Shah V, Atenafu E, Katz J. Influence of repeated painful procedures and sucrose analgesia on the development of hyperalgesia in newborn infants. Pain. 2009 Jul;144(1-2):43-8. doi: 10.1016/j.pain.2009.02.012. Epub 2009 Mar 28. PMID 19329255
- [Background] Jacobson RM, Swan A, Adegbenro A, Ludington SL, Wollan PC, Poland GA; Vaccine Research Group. Making vaccines more acceptable--methods to prevent and minimize pain and other common adverse events associated with vaccines. Vaccine. 2001 Mar 21;19(17-19):2418-27. doi: 10.1016/s0264-410x(00)00466-7. PMID 11257372
- [Background] Reis EC. Multiple scheduled injections contribute to missed opportunities to immunize during well care visits. Ambul Child Health 1997;3:172
- [Background] Woodin KA, Rodewald LE, Humiston SG, Carges MS, Schaffer SJ, Szilagyi PG. Physician and parent opinions. Are children becoming pincushions from immunizations? Arch Pediatr Adolesc Med. 1995 Aug;149(8):845-9. doi: 10.1001/archpedi.1995.02170210019003. PMID 7633536
- [Background] Shah V, Taddio A, Ohlsson A. Randomised controlled trial of paracetamol for heel prick pain in neonates. Arch Dis Child Fetal Neonatal Ed. 1998 Nov;79(3):F209-11. doi: 10.1136/fn.79.3.f209. PMID 10194994
- [Background] Howard CR, Howard FM, Weitzman ML. Acetaminophen analgesia in neonatal circumcision: the effect on pain. Pediatrics. 1994 Apr;93(4):641-6. PMID 8134222
- [Background] Taddio A, Manley J, Potash L, Ipp M, Sgro M, Shah V. Routine immunization practices: use of topical anesthetics and oral analgesics. Pediatrics. 2007 Sep;120(3):e637-43. doi: 10.1542/peds.2006-3351. PMID 17766503
- [Background] Prymula R, Siegrist CA, Chlibek R, Zemlickova H, Vackova M, Smetana J, Lommel P, Kaliskova E, Borys D, Schuerman L. Effect of prophylactic paracetamol administration at time of vaccination on febrile reactions and antibody responses in children: two open-label, randomised controlled trials. Lancet. 2009 Oct 17;374(9698):1339-50. doi: 10.1016/S0140-6736(09)61208-3. PMID 19837254
- [Background] Stevens B, Yamada J, Ohlsson A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD001069. doi: 10.1002/14651858.CD001069.pub3. PMID 20091512
- [Background] Harrison D, Bueno M, Yamada J, Adams-Webber T, Stevens B. Analgesic effects of sweet-tasting solutions for infants: current state of equipoise. Pediatrics. 2010 Nov;126(5):894-902. doi: 10.1542/peds.2010-1593. Epub 2010 Oct 11. PMID 20937658
- [Background] Bo LK, Callaghan P. Soothing pain-elicited distress in Chinese neonates. Pediatrics. 2000 Apr;105(4):E49. doi: 10.1542/peds.105.4.e49. PMID 10742370
- [Background] Field T, Goldson E. Pacifying effects of nonnutritive sucking on term and preterm neonates during heelstick procedures. Pediatrics. 1984 Dec;74(6):1012-5. PMID 6504620
- [Background] Leite AM, Linhares MB, Lander J, Castral TC, dos Santos CB, Silvan Scochi CG. Effects of breastfeeding on pain relief in full-term newborns. Clin J Pain. 2009 Nov-Dec;25(9):827-32. doi: 10.1097/AJP.0b013e3181b51191. PMID 19851165
- [Background] Gray L, Miller LW, Philipp BL, Blass EM. Breastfeeding is analgesic in healthy newborns. Pediatrics. 2002 Apr;109(4):590-3. doi: 10.1542/peds.109.4.590. PMID 11927701
- [Background] Gray L, Watt L, Blass EM. Skin-to-skin contact is analgesic in healthy newborns. Pediatrics. 2000 Jan;105(1):e14. doi: 10.1542/peds.105.1.e14. PMID 10617751
- [Background] Prasopkittikun T, Tilokskulchai F. Management of pain from heel stick in neonates: an analysis of research conducted in Thailand. J Perinat Neonatal Nurs. 2003 Oct-Nov;17(4):304-12. doi: 10.1097/00005237-200310000-00009. PMID 14655790
- [Background] Campos RG. Soothing pain-elicited distress in infants with swaddling and pacifiers. Child Dev. 1989 Aug;60(4):781-92. PMID 2758876
- [Background] O'Sullivan A, O'Connor M, Brosnahan D, McCreery K, Dempsey EM. Sweeten, soother and swaddle for retinopathy of prematurity screening: a randomised placebo controlled trial. Arch Dis Child Fetal Neonatal Ed. 2010 Nov;95(6):F419-22. doi: 10.1136/adc.2009.180943. Epub 2010 Sep 28. PMID 20876596
- [Background] Karp, Harvey. The Happiest Baby on the Block. New York, NY: Bantam Books; 2003
- [Background] Taddio A, Ilersich AL, Ipp M, Kikuta A, Shah V; HELPinKIDS Team. Physical interventions and injection techniques for reducing injection pain during routine childhood immunizations: systematic review of randomized controlled trials and quasi-randomized controlled trials. Clin Ther. 2009;31 Suppl 2:S48-76. doi: 10.1016/j.clinthera.2009.07.024. PMID 19781436
- [Background] Schade JG, Joyce BA, Gerkensmeyer J, Keck JF. Comparison of three preverbal scales for postoperative pain assessment in a diverse pediatric sample. J Pain Symptom Manage. 1996 Dec;12(6):348-59. doi: 10.1016/s0885-3924(96)00182-0. PMID 8973044
- [Background] McGrath PA. Pain in Children: Nature, Assessment, and Treatment. New York, NY:Guilford Press;1990.
- [Background] Blass EM. Milk-induced hypoalgesia in human newborns. Pediatrics. 1997 Jun;99(6):825-9. doi: 10.1542/peds.99.6.825. PMID 9164777
- [Background] Liu Y, von Deneen KM, Kobeissy FH, Gold MS. Food addiction and obesity: evidence from bench to bedside. J Psychoactive Drugs. 2010 Jun;42(2):133-45. doi: 10.1080/02791072.2010.10400686. PMID 20648909
- [Background] Berthoud HR, Lenard NR, Shin AC. Food reward, hyperphagia, and obesity. Am J Physiol Regul Integr Comp Physiol. 2011 Jun;300(6):R1266-77. doi: 10.1152/ajpregu.00028.2011. Epub 2011 Mar 16. PMID 21411768
- [Background] Stice E, Yokum S, Burger KS, Epstein LH, Small DM. Youth at risk for obesity show greater activation of striatal and somatosensory regions to food. J Neurosci. 2011 Mar 23;31(12):4360-6. doi: 10.1523/JNEUROSCI.6604-10.2011. PMID 21430137
- [Background] Pickering, LK, ed. RedBook: 2009 Report of the Committee on Infectious Diseases. 28th ed. Elk Grove Village, IL: American Academy of Pediatrics; 2009
- [Background] Tuck RH. Coding and payment for immunizations. Pediatr Ann. 2006 Jul;35(7):507-12. doi: 10.3928/0090-4481-20060701-07. PMID 16895151
- [Derived] Harrington JW, Logan S, Harwell C, Gardner J, Swingle J, McGuire E, Santos R. Effective analgesia using physical interventions for infant immunizations. Pediatrics. 2012 May;129(5):815-22. doi: 10.1542/peds.2011-1607. Epub 2012 Apr 16. PMID 22508924
- See also: Demonstration of the 5 S's — http://www.youtube.com/watch?v=WkR_e1L6zxI)